CLINICAL TRIAL: NCT05465382
Title: The Effect of Early Saline Lavage on Synovial Fluid Composition Following Human Intra-Articular Ankle Fracture
Brief Title: Intra Articular Ankle Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00110537
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Intra-Articular Fractures
MeSH Terms: conditions — Intra-Articular Fractures

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of two groups: 1) intra-articular saline lavage, vs 2) no intra-articular saline lavage. Intra-articular aspiration of synovial fluid from the injured ankle will occur both at the time of presentation to the emergency department and at the time of surgery.
Who Masked: Participant
Masking Description: Randomization will occur by the opening of pre-prepared envelopes which will be stored in the orthopaedic resident office. Envelopes will be labeled #1-#60. Thirty envelopes will contain a note card labeled "Group 1" and Thirty envelopes will contain a note card labeled "Group 2". Envelopes will be pre-prepared by key study personnel not involved in the consent or randomization process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intra-articular saline lavage (Experimental): Subjects in Group 1 will then undergo saline joint lavage as follows:
  Subjects will undergo aspiration of the injured ankle joint via the standard anteromedial arthroscopy portal approach. This will be performed with sterile technique using a 16-gauge needle attached to a 10cc syringe. After synovial fluid aspiration, three 10cc syringes will be filled with 10cc of sterile 0.9% normal saline. Normal saline will be injected into the ankle joint and withdrawn from the joint via the existing anteromedial 16 gauge needle. After three rounds of lavage, 10cc of 1% lidocaine without epinephrine will be injected into the joint via the existing anteromedial 16-gauge needle. Subjects will undergo a period of soft tissue rest to allow for the resolution of soft tissue swelling. At the time of surgical fixation subjects will again undergo intra-articular aspiration of the injured ankle joint.
  Interventions: Device: Saline Lavage; Drug: Lidocaine - intra-articular injection; Other: Synovial Fluid Aspiration
- No intra-articular saline lavage (Active Comparator): Subjects in group 2 will not undergo normal saline lavage.
  Interventions: Other: No intra-articular saline lavage; Drug: Lidocaine - intra-articular injection; Other: Synovial Fluid Aspiration

INTERVENTIONS:
Device: Saline Lavage — Three rounds of 10cc of sterile 0.9% normal saline will be injected into the injured ankle joint and withdrawn from the joint using an anteromedial 16-gauge needle attached to a 10cc syringe.
  Arms: Intra-articular saline lavage
Other: No intra-articular saline lavage — Subjects in group 2 will not undergo normal saline lavage.
  Arms: No intra-articular saline lavage
Drug: Lidocaine - intra-articular injection — Intra-articular injection of 10cc of 1% lidocaine without epinephrine via the existing anteromedial 16-gauge needle.
Other: Synovial Fluid Aspiration — Aspiration of ankle joint via standard anteromedial approach. Performed using sterile technique using 16-guage needle attached to 10cc syringe.

SUMMARY:
The purpose of this study is to examine the effect of early, percutaneous, intra-articular saline lavage on the undiluted synovial fluid microenvironment during the acute phase following intra-articular fracture of the human ankle. We hypothesize that early intervention with percutaneous joint lavage in the first 0-48 hours after injury will attenuate the production of pro-inflammatory cytokines, MMP's and cartilage breakdown products compared to non-lavaged control subjects at the time of surgical fixation.

DETAILED DESCRIPTION:
Saline joint lavage represents a potentially simple, low-risk and minimal-cost intervention which has not been previously studied for the purpose of reducing the post-fracture inflammatory burden in human subjects. Open joint lavage at the time of definitive surgical fixation is within the standard of care, but typically occurs greater than 10 days after injury by which time cartilage degradation has already begun. Early, saline lavage during initial presentation to the emergency department may theoretically alter the progression of the intra-articular inflammatory response by evacuating the bulk of the developing synovial-fluid fracture hematoma.

The vast majority of ankle fractures present to the ER or urgent care within a day of fracture. Moreover, a large subset of these fractures require reduction (fracture setting) that is painful. It is our standard of care to perform an intra-articular lidocaine injection before reduction. We will take advantage of this standard of care needle insertion to the fractured ankle to perform saline joint lavage to diminish this early inflammatory burden. Adult patients presenting to the Duke University Hospital Emergency Department with an intra-articular fracture of the ankle joint between 0-48 hours from the time of injury will be eligible for inclusion. Patients will be randomized into one of two groups: 1) intra-articular saline lavage, vs 2) no intra-articular saline lavage. Intra-articular aspiration of synovial fluid from the injured ankle will occur both at the time of presentation to the emergency department and at the time of surgery. These synovial fluid samples will be analyzed for differences in key pro-inflammatory cytokines, matrix metalloproteinases and cartilage breakdown products to determine if early saline lavage effects the composition of the synovial fluid micro-environment.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (over 18 years of age)
* Must be treated at Duke University Hospital Emergency Department
* Intra-articular fracture of the ankle joint (any fracture of the fibula or tibia in which the fracture line(s) exit into the cartilage surface of the ankle joint)
* Subjects presenting between 0-48 hours from the time of injury

Exclusion Criteria:

* Age < 18 y.o.
* Open fracture
* Nonoperatively treated fractures
* Subjects presenting >48 hours from the time of injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Change in cytokines levels at specific time points after injury | baseline, in the OR after anesthesia is induced (generally within 24 hours of lavage), and 1 to 2 weeks post-injury.
  Analyte concentrations will be collected during standardized aspirations at the time of emergency department presentation and at the time of surgery.
Change in matrix metalloproteinase levels at specific time points after injury | baseline, in the OR after anesthesia is induced (generally within 24 hours of lavage), and 1 to 2 weeks post-injury.
  Analyte concentrations will be collected during standardized aspirations at the time of emergency department presentation and at the time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Adams, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huch K, Kuettner KE, Dieppe P. Osteoarthritis in ankle and knee joints. Semin Arthritis Rheum. 1997 Feb;26(4):667-74. doi: 10.1016/s0049-0172(97)80002-9. PMID 9062947
- [Background] Brown TD, Johnston RC, Saltzman CL, Marsh JL, Buckwalter JA. Posttraumatic osteoarthritis: a first estimate of incidence, prevalence, and burden of disease. J Orthop Trauma. 2006 Nov-Dec;20(10):739-44. doi: 10.1097/01.bot.0000246468.80635.ef. PMID 17106388
- [Background] Delco ML, Kennedy JG, Bonassar LJ, Fortier LA. Post-traumatic osteoarthritis of the ankle: A distinct clinical entity requiring new research approaches. J Orthop Res. 2017 Mar;35(3):440-453. doi: 10.1002/jor.23462. Epub 2016 Nov 8. PMID 27764893
- [Background] Buckwalter JA, Brown TD. Joint injury, repair, and remodeling: roles in post-traumatic osteoarthritis. Clin Orthop Relat Res. 2004 Jun;(423):7-16. PMID 15232420
- [Background] McKinley TO, Tochigi Y, Rudert MJ, Brown TD. The effect of incongruity and instability on contact stress directional gradients in human cadaveric ankles. Osteoarthritis Cartilage. 2008 Nov;16(11):1363-9. doi: 10.1016/j.joca.2008.04.005. Epub 2008 Jun 3. PMID 18511308
- [Background] Dirschl DR, Marsh JL, Buckwalter JA, Gelberman R, Olson SA, Brown TD, Llinias A. Articular fractures. J Am Acad Orthop Surg. 2004 Nov-Dec;12(6):416-23. doi: 10.5435/00124635-200411000-00006. PMID 15615507
- [Background] Giannoudis PV, Tzioupis C, Papathanassopoulos A, Obakponovwe O, Roberts C. Articular step-off and risk of post-traumatic osteoarthritis. Evidence today. Injury. 2010 Oct;41(10):986-95. doi: 10.1016/j.injury.2010.08.003. PMID 20728882
- [Background] Allen NB, Abar B, Danilkowicz RM, Kraus VB, Olson SA, Adams SB. Intra-Articular Synovial Fluid With Hematoma After Ankle Fracture Promotes Cartilage Damage In Vitro Partially Attenuated by Anti-Inflammatory Agents. Foot Ankle Int. 2022 Mar;43(3):426-438. doi: 10.1177/10711007211046952. Epub 2021 Oct 7. PMID 34617803
- [Background] Hembree WC, Ward BD, Furman BD, Zura RD, Nichols LA, Guilak F, Olson SA. Viability and apoptosis of human chondrocytes in osteochondral fragments following joint trauma. J Bone Joint Surg Br. 2007 Oct;89(10):1388-95. doi: 10.1302/0301-620X.89B10.18907. PMID 17957084
- [Background] Adams SB, Setton LA, Bell RD, Easley ME, Huebner JL, Stabler T, Kraus VB, Leimer EM, Olson SA, Nettles DL. Inflammatory Cytokines and Matrix Metalloproteinases in the Synovial Fluid After Intra-articular Ankle Fracture. Foot Ankle Int. 2015 Nov;36(11):1264-71. doi: 10.1177/1071100715611176. Epub 2015 Oct 8. PMID 26449389
- [Background] Adams SB, Reilly RM, Huebner JL, Kraus VB, Nettles DL. Time-Dependent Effects on Synovial Fluid Composition During the Acute Phase of Human Intra-articular Ankle Fracture. Foot Ankle Int. 2017 Oct;38(10):1055-1063. doi: 10.1177/1071100717728234. Epub 2017 Sep 11. PMID 28891711
- [Background] Kimmerling KA, Furman BD, Mangiapani DS, Moverman MA, Sinclair SM, Huebner JL, Chilkoti A, Kraus VB, Setton LA, Guilak F, Olson SA. Sustained intra-articular delivery of IL-1RA from a thermally-responsive elastin-like polypeptide as a therapy for post-traumatic arthritis. Eur Cell Mater. 2015 Jan 31;29:124-39; discussion 139-40. doi: 10.22203/ecm.v029a10. PMID 25636786
- [Background] Furman BD, Mangiapani DS, Zeitler E, Bailey KN, Horne PH, Huebner JL, Kraus VB, Guilak F, Olson SA. Targeting pro-inflammatory cytokines following joint injury: acute intra-articular inhibition of interleukin-1 following knee injury prevents post-traumatic arthritis. Arthritis Res Ther. 2014 Jun 25;16(3):R134. doi: 10.1186/ar4591. PMID 24964765